CLINICAL TRIAL: NCT01083498
Title: Ablative Fractional Laser Therapy as Treatment for Becker's Nevus; a Pilot Study
Brief Title: Fractional Laser as Treatment Option for Various Pigment Disorders
Acronym: fractional-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Netherlands Institute for Pigment Disorders (Other)
Responsible Party: A Wolkerstorfer, MD PhD, Netherlands Institute for Pigment Disorders
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: fractional-2
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Pigmentation Disorder
Keywords: Becker's nevus; ablative fractional laser therapy; randomized controlled trial; split-lesion design
MeSH Terms: conditions — Pigmentation Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ablative fractional laser (Experimental): In each patient, a square test region of 5-10 cm2 was treated with ablative fractional laser in three sessions in combination with intermittent topical bleaching with triple topical therapy (hydroquinone 5%, tretinoin 0.05%, triamcinolone acetonide 0.1% cream) to prevent laser-induced postinflammatory hyperpigmentation.
  Note: this study had a split-lesion design. In each patient, two test regions were randomized to receive either ablative fractional laser therapy or no treatment.
  Interventions: Device: Ablative fractional laser therapy
- Control (No Intervention): In each patient, a square test region of 5-10 cm2 was treated with topical bleaching with triple topical therapy (hydroquinone 5%, tretinoin 0.05%, triamcinolone acetonide 0.1% cream)alone (to allow comparison of the regions).
  Note: this study had a split-lesion design. In each patient, two test regions were randomized to receive either ablative fractional laser therapy or no treatment.

INTERVENTIONS:
Device: Ablative fractional laser therapy — 10,600 nm ablative fractional laser Irradiance: 10 mJ/microbeam. Coverage: 35-45%. Number of treatment sessions: 3
  Other Names: Fraxel re:pair, Solta Medical Inc., Hayward, CA
  Arms: Ablative fractional laser

SUMMARY:
The purpose of this study is to determine whether the use of ablative fractional laser is effective in the treatment of Becker's nevus.

DETAILED DESCRIPTION:
Becker's nevus (BN) is an uncommon pigment disorder of the epidermis characterized by increased pigmentation, a slightly elevated, verrucous surface of the affected skin and sometimes hyperpigmentation. No effective treatment is available. Several laser modalities have been applied in the treatment of Becker's nevus in uncontrolled studies with varying results. Recently, fractional laser therapy was suggested as treatment option for Becker's nevus. In fractional laser therapy, microscopic columns of skin are coagulated or ablated, leaving the surrounding tissue intact, which enhances healing of the treated skin. In this study, the efficacy and safety of ablative fractional laser therapy was assessed in the treatment of Becker's nevus.

ELIGIBILITY:
Inclusion Criteria:

* Becker nevus
* Subjects attending the outpatient department of the Netherlands Institute for Pigment Disorders
* Age at least 18 years
* Subject is willing and able to give written informed consent

Exclusion Criteria:

* use of bleaching creams during the past six weeks
* history of keloid
* active eczema
* suspected hypersensitivity to lidocaine or triple therapy
* use of isotretinoin in the past six months
* high exposure of the lesion to sunlight or UV light (UVA or UVB).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Physician's global assessment | T0, 3 and 6 months follow-up
  Improvement of hyperpigmentation was assessed by an independent blinded dermatologist. The results were scored on a scale from zero to six (0: total clearance (100% improvement), 1: almost total clearance (90-99% improvement), 2: distinct clearance (75-89% improvement) 3: moderate clearance (50-74% improvement) 4: mild clearance (25-49% improvement) 5: no change, 6: worsening of hyperpigmentation).

SECONDARY OUTCOMES:
L-value | T0, 3 and six months follow-up
  Improvement of hyperpigmentation was assessed by color measurement through reflectance spectroscopy (Microflash 200 d, Datacolor International, Lawrenceville, GA). This instrument, with an aperture of 4 mm, determines color by measuring the intensity of reflected light of particular wavelengths. In this study, the obtained L value, reflecting the lightness of the measured area of skin, was used.
Melanin index | T0, 3 and 6 months follow-up
  Melanin index was measured using a spectrometer (Derma-Spectrometer, Cortex Technology ApS, Hadsund, Denmark) in order to assess changes in the amount of dermal and epidermal melanin.
Patient's global assessment | 3 and 6 months follow-up
  Patients were asked to score the improvement of hyperpigmentation on a visual analogue scale (VAS) from 0 to 10 (Patient's Global Assessment, PGA) at all follow-up moments.
Patient's satisfaction | 3 and 6 months follow-up
  Patient's satisfaction was scored on a visual analogue scale (VAS) from 0 to 10.
Histopathologic assessment | 3 months follow-up
  In order to evaluate for microscopic and ultrastructural treatment induced changes, 2 mm punch biopsies were taken from all patients at three months follow-up. Biopsies were taken from the optical centre of both treated and control site. All biopsy specimens were split for processing for light microscopy. .... was assessed by an independent blinded pathologist.